CLINICAL TRIAL: NCT07161362
Title: Measurement of Utilization of Dental Care and Dental Services Provided in Pediatric Dentistry Department at El Kasr El Einy : Longitudinal Observational Study
Brief Title: Measurement of Dental Health Care Utilization
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ola Emad, M. D. candidate, Kasr El Aini Hospital
Other Study IDs: CU311032
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2023-01

CONDITIONS: Utilization of Dental Care

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
measurement of utilization of dental services in pediatric department in faculty of dentistry in Cairo University within 18 month starting from January 2023 till June 2024 depending on recorded data.

ELIGIBILITY:
Inclusion Criteria:

* each patient available records

Exclusion Criteria:

* if records is not available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: records of patients present in pediatric department in faculty of dentistry in Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 1059 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Measurement of utilization of dental care of each service in percentage according to total services. | 18 months from Jan 2023 to June 2024

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry at Cairo University, Cairo, Egypt